CLINICAL TRIAL: NCT02682186
Title: Effects of the Pectoral Blocks in the Prosthetic Breast Expansion Surgery : Prospective, Randomized, Double Blind Study.
Brief Title: Pectoral Nerve Block for Analgesia After Breast Augmentation
Acronym: PECS B&BS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 95832; 2015-002368-17 (EudraCT Number)
Record Dates: First submitted 2016-02-04; First posted 2016-02-15 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Ambulatory Plastic Surgery; Esthetic Prosthetic Breast Expansion
Keywords: Prosthetic breast surgery; Locoregional anesthesia; Pectoral nerve block; Pain; Postoperative analgesia
MeSH Terms: conditions — Pain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (1) (No Intervention): The PECS Blocks are not (1) performed.
- PECS group (2) (Experimental): The PECS Blocks are performed (2): A single injection of Ropivacaine after dilution with sodium chloride 0.9% per fascial plane and per side.
  Interventions: Drug: Ropivacaine after dilution with sodium chloride 0.9%

INTERVENTIONS:
Drug: Ropivacaine after dilution with sodium chloride 0.9% — After the anesthesic induction, the interventional team composed by at least a senior anaesthesiologist and a nurse anesthestic, will survey the patient and perform the Pecs blocks, whereas the anesthetic team is outside the room.
  Realization of Pecs blocks 1 and 2 : the patient is in supine position with placing the upper limb in abduction position, a 100 mm needle is inserted under ultrasound using a linear US probe of high frequency after sheathing.
  In the other group, sterilization, sheating and US are performed but the needle is not inserted.
  Arms: PECS group (2)

SUMMARY:
Breast augmentation is among the most popular surgical procedures performed in the world with approximately 1,773,584 performed in 2013. This surgical intervention generates important pains during postsurgical recovery. A multimodal analgesia, based on the recommendations is proposed to the patients .The pectoral nerve block is an innovative technique of locoregional anesthesia that has already been successfully used in breast surgery. Its realization is fast, simple, and it would be superior compared with a paravertebral block within the framework of mastectomy. The interest of this technique has never been assessed in esthetic breast surgery. The aim of this study is to evaluate the analgesic efficacy of the association of " Pecs blocks 1 and 2 " on pain intensity after breast augmentation surgery.

DETAILED DESCRIPTION:
The investigators hypothesized that the "Pecs blocks 1 and 2" will provide a decrease of the maximal pain of the first 6 post-operative hours after prosthetic breast expansion. The pain will be assessed according to a numerical scale. This prospective, randomized, double blind study will include 92 patients successively during two years, randomized into two arms : Pecs group and Control group, which will respectively have the block, and no block. The rest of the anesthesic and surgical care will be identical.

An intervention team (which will be different from the anesthesic team), will be alone with the patient for 15 minutes, and will realize or not the Pecs blocks according to the previous randomisation so that all caregivers taking in charge the patients as well as research observers will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to a national insurance scheme
* Having signed the informed consent for this study
* Score of American Society of Anesthesiology ( ASA) 1-3
* Be hospitalized in the ambulatory care unit (UCA) or plastic surgery service for a scheduled esthetic prosthetic breast expansion surgery.

Exclusion Criteria:

* Protected minor or major patients or in the incapacity to give his consent according to the article L1121-8 of the Code of the Health Public.
* Pregnant or breast-feeding women according to French law.
* Vulnerable people.
* Patients participating in another research
* Allergy with local anesthetics.
* Severe coagulopathy.
* Chronic painful Patients (long-term treatment by analgesics)
* Contraindication to use analgesics of the protocol.
* Change of breast prostheses

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Maximal value of pain intensity according to the numerical scale within the six first hours | up to First six postoperative hours

SECONDARY OUTCOMES:
Maximal value of the pain at day 1 and until day 5 | Five days
  Value of pain according to a Numeric scale , recorded at day 1 in the hospital, and until day five by phone interview.
Morphinics side effects such as nausea / vomiting, constipation, pruritus; analgesic consumption, surgical complication, satisfaction questionaire | Five days
  Any of side effect

CONTACTS AND LOCATIONS:
Overall Officials: Gérald GC CHANQUES, MD, PhD, Study Chair — Montpellier University Hospital
Locations (3):
- France (3):
  - UH Montpellier - Hôpital Gui de Chauliac, Montpellier
  - UH Montpellier, Montpellier
  - CHU Nîmes, Nîmes

IPD SHARING:
Plan to Share IPD: Undecided